CLINICAL TRIAL: NCT06437548
Title: Spinal Cord Stimulation for Reanimation After Nervous System Injury
Brief Title: Epidural Stimulation for Upper Extremity Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, MD PhD, Director of Neurosurgical Trauma, Associate Professor of Neurosurgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P000185
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injury Cervical; Tetraplegia
Keywords: spinal; cord; stimulation; percutaneous; peripheral; nerve; transfer
MeSH Terms: conditions — Quadriplegia; Cone-Rod Dystrophies

STUDY DESIGN:
Intervention Model Description: Percutaneous temporary spinal cord stimulator. Parameters for upper extremity motor function will be assessed with the stimulation turned on and off. Muscle strength and force will be assessed with the stim turned on and off.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Percutaneous spinal cord stimulation (Experimental): All participants will undergo baseline muscle strength and force assessments. Participants will also answer questionnaires on pain and quality of life. An optional nerve health assessment with needle electromyography and neuroimaging may be performed.
  Participants will undergo clinically indicated percutaneous (temporal) cervical epidural leads placement.
  Weeks 0-4 post-leads placement: during weekly visits upper extremity muscle strength and force will be assessed, pain and quality of life questionnaires will be completed (1 research visit per week)
  At approximately 28 days temporary leads will be removed.
  At the last visit, muscle strength and force in upper extremity muscle groups will be assessed, participants will complete pain and quality of life questionnaires. Participants may choose to undergo an optional nerve health assessment with needle electromyography and neuroimaging.
  Interventions: Device: Percutaneous spinal cord stimulation

INTERVENTIONS:
Device: Percutaneous spinal cord stimulation — The parameters of percutaneous cervical spinal cord stimulation leads will be adjusted for optimal upper extremity motor function.

SUMMARY:
Restoring upper extremity function in patients with cervical spinal cord injury is extremely important for patients' independence and quality of life.

At present, there are limited options for hand or arm reanimation in this patient population. Nerve transfer is one such option that can partially restore the natural movement of hand or arm function in select patients.

The investigators are interested in understanding whether recovery of hand or arm motor function after nerve transfer can be augmented by cervical epidural spinal cord stimulation.

DETAILED DESCRIPTION:
The study will enroll up to 20 participants in a single arm prospective clinical study. Potential participants will have already had a nerve transfer surgery more than 6 months prior to enrollment and will have also completed post-nerve transfer physical /occupational neurorehabilitation.

At baseline, upper extremity muscle strength, muscle force and nerve health with needle electromyography and neuroimaging will be tested.

Patients will undergo percutaneous (temporary) spinal cord stimulator leads placement in the cervical supralesional spine region.

Week 0-4: Weekly testing of motor function and muscle contraction force with the stimulation turned on versus turned off will be performed. Stimulation parameters for each target upper extremity muscle will also be documented.

Temporary leads will be removed after approximately 4 weeks.

At the last research visit at approximately 6-7 weeks post leads placement muscle strength/force will be assessed to determine the duration of the stimulation effect (if it is sustained). To assess any improvement of nerve health, neuroimaging and electromyography will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤65
* Provides informed consent
* History of upper extremity nerve transfer > 6 months prior to enrollment
* Completion of standard post-nerve transfer occupational therapy
* Baseline upper extremity strength of < 5/5 grade with the MRC
* Scheduled to undergo a cervical spinal cord stimulation procedure for chronic pain refractory to first line therapy
* Willing and able to adhere to the study protocol

Exclusion Criteria:

* Central nervous system (CNS) malignancy
* A contraindication to the SCS procedure
* Diagnosis that precludes the patient from full participation in the protocol
* A functional implanted device (pacemaker, vagus nerve device, baclofen pump)
* Botulinum toxin injection in upper extremity muscles < 6 months prior to enrollment
* For female participants, current/planned pregnancy (females of childbearing age will be asked to take a pregnancy test on the day of the intervention)
* Other factors that prevent participation in the opinion of the surgeon-principal investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Nerve transfer recipient muscle strength | 0-6 weeks
  Change in Medical Research Council (MRC) grade of recipient nerve transfer muscle group with spinal cord stimulation activated. MRC ranges from 0 (no visible muscle contraction) to 5 (normal muscle strength against full resistance). A larger number represents a better outcome.

SECONDARY OUTCOMES:
Nerve transfer recipient muscle force | 0-6 weeks
  Change in muscle force generated by recipient nerve transfer muscle group with spinal cord stimulation activated. Muscle force is measured with a hand-held dynamometer. This is measured in Newtons, with a larger number meaning greater force and a better outcome.
Neck and upper extremity pain | 0-6 weeks
  Change in neck and upper extremity pain measured with the Numeric Rating Scale (NRS). NRS scale ranges from 0 (No pain) to 10 (worst possible pain), with a lower number representing a better outcome. A positive change in NRS from baseline to follow-up visits suggests improvement of pain.
Amplitude of percutaneous stimulation | 0-4 weeks
  Optimized amplitude of percutaneous stimulation for each upper extremity muscle for voluntary hand/arm motor function will be documented. Amplitude is measured in miliAmperes.
Frequency of percutaneous stimulation | 0-4 weeks
  Optimized frequency of percutaneous stimulation for each upper extremity muscle for voluntary hand/arm motor function will be documented. Frequency is measured in Hz (Hertz).
Pulse width of percutaneous stimulation | 0-4 weeks
  Optimized pulse width of percutaneous stimulation for each upper extremity muscle for voluntary hand/arm motor function will be documented. Pulse width is measured in microseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, MD PhD, Study Chair — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside of the study, except as required de-identified data for publication purposes.

REFERENCES:
- [Background] Bertelli JA, Ghizoni MF. Nerve transfers for restoration of finger flexion in patients with tetraplegia. J Neurosurg Spine. 2017 Jan;26(1):55-61. doi: 10.3171/2016.5.SPINE151544. Epub 2016 Aug 5. PMID 27494781
- [Background] Fox IK. Nerve Transfers in Tetraplegia. Hand Clin. 2016 May;32(2):227-42. doi: 10.1016/j.hcl.2015.12.013. Epub 2016 Mar 10. PMID 27094894
- [Background] Lu DC, Edgerton VR, Modaber M, AuYong N, Morikawa E, Zdunowski S, Sarino ME, Sarrafzadeh M, Nuwer MR, Roy RR, Gerasimenko Y. Engaging Cervical Spinal Cord Networks to Reenable Volitional Control of Hand Function in Tetraplegic Patients. Neurorehabil Neural Repair. 2016 Nov;30(10):951-962. doi: 10.1177/1545968316644344. Epub 2016 May 18. PMID 27198185
- [Background] Barra B, Conti S, Perich MG, Zhuang K, Schiavone G, Fallegger F, Galan K, James ND, Barraud Q, Delacombaz M, Kaeser M, Rouiller EM, Milekovic T, Lacour S, Bloch J, Courtine G, Capogrosso M. Epidural electrical stimulation of the cervical dorsal roots restores voluntary upper limb control in paralyzed monkeys. Nat Neurosci. 2022 Jul;25(7):924-934. doi: 10.1038/s41593-022-01106-5. Epub 2022 Jun 30. PMID 35773543
- [Background] Greiner N, Barra B, Schiavone G, Lorach H, James N, Conti S, Kaeser M, Fallegger F, Borgognon S, Lacour S, Bloch J, Courtine G, Capogrosso M. Recruitment of upper-limb motoneurons with epidural electrical stimulation of the cervical spinal cord. Nat Commun. 2021 Jan 19;12(1):435. doi: 10.1038/s41467-020-20703-1. PMID 33469022
- [Background] Powell MP, Verma N, Sorensen E, Carranza E, Boos A, Fields DP, Roy S, Ensel S, Barra B, Balzer J, Goldsmith J, Friedlander RM, Wittenberg GF, Fisher LE, Krakauer JW, Gerszten PC, Pirondini E, Weber DJ, Capogrosso M. Epidural stimulation of the cervical spinal cord for post-stroke upper-limb paresis. Nat Med. 2023 Mar;29(3):689-699. doi: 10.1038/s41591-022-02202-6. Epub 2023 Feb 20. PMID 36807682